CLINICAL TRIAL: NCT04872595
Title: Phase 2 Study of Personalized r-ATG Dosing to Improve Survival Through Enhanced Immune Reconstitution in Pediatric and Adult Patients Undergoing Ex-vivo CD34-Selected Allogeneic-HCT (PRAISE-IR)
Brief Title: A Modified Dose of Rabbit Anti-thymocyte Globulin (rATG) in Children and Adults Receiving Treatment to Help Prepare Their Bodies for a Bone Marrow Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-193
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoid Leukemia (ALL); Myelodysplastic Syndromes (MDS)
Keywords: personalized rabbit ATG (P-rATG); ex-vivo CD34+ T cell depleted; total body irradiation; thiotepa; cyclophosphamide; busulfan; melphalan; fludarabine; 21-193
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — Thiotepa; Cyclophosphamide; Busulfan; Melphalan; fludarabine

STUDY DESIGN:
Intervention Model Description: This phase 2 study is to assess the effects of personalized rabbit ATG (P-rATG) dosing on CD4+ immune reconstitution (CD4+IR) based on a pharmacokinetic/pharmacodynamic (PK/PD) model in patients with hematologic malignancies undergoing peripheral blood mobilized, ex-vivo CD34+ T cell depleted, allogeneic, hematopoietic cell transplantation (CD34+/TCD allo-HCT)1.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- P-rATG with total body irradiation, thiotepa, cyclophosphamide (Experimental): P-rATG days (always starting on Day -12 to -10)
  * Hyper fractionated total body irradiation (1375 - 1500cGy*) Day -9 to -6
  * Thiotepa (5mg/kg/day x 2 day) Day -5 to -4
  * Cyclophosphamide (60mg/kg/day x 2 days) Day -3 to -2
  * GCSF Day +7 *TBI dose in 125cGy fractions (with lung shielding) and total dose to be determined by treating physician/radiation oncology and is based off age, stage of disease, and anesthesia requirements.
  Interventions: Other: Personalized rATG (P-rATG); Radiation: Hyper fractionated total body irradiation; Drug: Thiotepa; Drug: Cyclophosphamide; Drug: GCSF
- P-rATG with busulfan, melphalan and fludarabine (Experimental): P-rATG days (Appendix A - always starting on Day -12 to -10)
  * Busulfan -Day -9 to -7
  * Initial dose per table in Appendix B; doses 2-3 to be adjusted per PK for target cumulative exposure of 65 mg*h/L Melphalan (70mg/m2/day x 2 days) Day -6 to -5
  * Fludarabine (25mg/m2/day x 5 days) Day -6 to -2
  * GCSF Day +7
  Interventions: Other: Personalized rATG (P-rATG); Drug: GCSF; Drug: Busulfan; Drug: Melphalan; Drug: Fludarabine

INTERVENTIONS:
Other: Personalized rATG (P-rATG) — P-rATG days (always starting on Day -12 to -10)
Radiation: Hyper fractionated total body irradiation — (1375 - 1500cGy*) Day -9 to -6
  *TBI dose in 125cGy fractions (with lung shielding) and total dose to be determined by treating physician/radiation oncology and is based off age, stage of disease, and anesthesia requirements.
  Arms: P-rATG with total body irradiation, thiotepa, cyclophosphamide
Drug: Thiotepa — (5mg/kg/day x 2 day) Day -5 to -4
  Arms: P-rATG with total body irradiation, thiotepa, cyclophosphamide
Drug: Cyclophosphamide — (60mg/kg/day x 2 days) Day -3 to -2
  Arms: P-rATG with total body irradiation, thiotepa, cyclophosphamide
Drug: GCSF — Day +7
Drug: Busulfan — Day -9 to -7 doses 2-3 to be adjusted per PK for target cumulative exposure of 65 mg*h/L
  Arms: P-rATG with busulfan, melphalan and fludarabine
Drug: Melphalan — (70mg/m2/day x 2 days) Day -6 to -5
  Arms: P-rATG with busulfan, melphalan and fludarabine
Drug: Fludarabine — (25mg/m2/day x 5 days) Day -6 to -2
  Arms: P-rATG with busulfan, melphalan and fludarabine

SUMMARY:
The purpose of this study is to see if conditioning regimens that include personalized rabbit ATG (P-rATG) help the immune system recover sooner and decrease the chances of transplant-related side effects. Participants in this study will be children and adults who have acute leukemia or myelodysplastic syndrome (MDS), and will receive a standard conditioning regimen to prepare the body for an allogeneic hematopoietic cell transplant (allo-HCT). The conditioning regimen will include r-ATG, one of two combinations of chemotherapy, and possibly total body irradiation (TBI).

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving first peripheral blood mobilized ex-vivo CD34-selected T cell depleted allo-HCT for the following hematologic malignant conditions:

  * Acute myeloid leukemia (AML) with intermediate or high-risk features in CR1 or Relapse AML in ≥ CR2.
  * Must have MRD <5% (flow cytometry, molecular and/or cytogenetics accepted).
  * Acute leukemias of ambiguous lineage in ≥ CR1.
  * Must have MRD <5% (flow cytometry, molecular and/or cytogenetics accepted).
  * Acute lymphoid leukemia (ALL) in CR1 with clinical, flow cytometric, or molecular features indicating a high risk for relapse, or ALL in ≥ CR2.
  * Adult Patients - recommended but not required to be MRDnegative (by flow cytometry, molecular and/or cytogenetics).
  * Pediatric Patients - Must be MRD-negative by flow cytometry, molecular and/or cytogenetics.
  * Myelodysplastic syndromes (MDS) with least one of the following:
  * Revised International Prognostic Scoring System risk score of intermediate or higher at the time of transplant evaluation.
  * Life-threatening cytopenia.
  * Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype.
  * Therapy related disease or disease evolving from other malignant processes.
* Able to tolerate cytoreduction
* Patients age:

  * Regimen A: 4 - 60 years
  * Regimen B - no age restriction
* Adequate organ function is required, defined as follows:

  * Hepatic: Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia. Patients with hyperbilirubinemia related to paroxysmal nocturnal hemoglobinuria or other hemolytic disorders are eligible with PI approval.
  * Hepatic: AST, ALT, and alkaline phosphatase < 2.5 times the upper limit of normal unless thought to be disease-related.
  * Renal: serum creatinine <1.5x normal for age. If serum creatinine is outside the normal range, then CrCl > 50 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.72m2) >30% of predicted normal for age.
* Normal GFR by Age

  * 1 week 40.6 + / - 14.8
  * 2 - 8 weeks 65.8 + / - 24.8

    °> 8 weeks 95.7 +/- 21.7
  * 2 - 12 years 133 +/- 27
  * 13 - 21 years (males) 140 +/- 30
  * 13 - 21 years (females) 126.0 + / - 22.0
* Cardiac: LVEF ≥ 50% by MUGA or resting echocardiogram.
* Pulmonary: Pulmonary function testing (FEV1 and corrected DLCO) ≥ 50% predicted (pediatric patients unable to complete PFTs will need oxygen saturation as recorded by pulse oximetry of ≥92% on room air).
* Adequate performance status:

  * Age ≥ 16 years: ECOG ≤ 1 or Karnofsky 70%
  * Age < 16 years: Lansky 70%
* Each patient must be willing to participate as a research subject and must sign an informed consent form or legal guardian with assent as appropriate.

Exclusion Criteria:

* Patients with active extramedullary disease.
* Patients with active central nervous system malignancy.
* Uncontrolled infection at the time of allo-HCT.
* Patients who have undergone previous allo-HCT.
* Patient seropositivity for HIV I/II and/or HTLV I/II.
* Females who are pregnant or breastfeeding.
* Patients unwilling to use contraception during the study period.
* Patient or parent or guardian unable to give informed consent or unable to comply with the treatment protocol including research tests.

Donor Inclusion Criteria:

* Related or Unrelated Donors:

  °8/8 HLA matched at A, B, C, and DRB1 loci, as tested by DNA analysis.
* Able to provide informed consent for the donation process per institutional standards.
* Meet standard criteria for donor collection (e.g. National Marrow Donor Program Guidelines or collecting center guidelines as approved by treating physician).
* Provide GSCF mobilized peripheral blood stem cells

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who achieve CD4+IR | within 100 days of HCT
  is defined at CD4+ > 50u/L at two consecutive measures within 100 days post allo-HCT.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  The duration of time between HCT and death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Curran, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Scordo M, Perales MA, Mauguen A, Lin A, Kunvarjee B, Paes Pena M, Mcavoy D, Nguyen LK, Hogan M, Chapman N, Bieler J, Cho C, Gyurkocza B, Harris AC, Spitzer B, O'Reilly RJ, Jakubowski AA, Lin RJ, Papadopoulos EB, Politikos I, Ponce DM, Shaffer BC, Shah GL, Tamari R, Giralt SA, Boelens JJ, Curran KJ. Model-based antithymocyte globulin dosing in ex vivo CD34+ selected allogeneic haematopoietic cell transplantation: a single-centre, single-arm, phase 2 study. Lancet Haematol. 2025 Dec;12(12):e956-e965. doi: 10.1016/S2352-3026(25)00293-5. PMID 41338864
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT04872595/ICF_000.pdf